CLINICAL TRIAL: NCT02930200
Title: Pilot Randomized Clinical Trial of an Automated Smartphone Based Smoking Cessation Treatment
Brief Title: Clinical Trial of an Automated Smartphone Based Smoking Cessation Treatment
Acronym: Smart-T2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7195
Record Dates: First submitted 2016-10-07; First posted 2016-10-12 (Estimated); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Smartphone Based Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment as Usual (Active Comparator): Behavioral: Treatment as Usual (TAU) is the Tobacco Treatment Research Program (TTRP) which offers all components of an intensive tobacco treatment intervention including: 1) initial assessment of willingness to participate, 2) the use of multiple types of clinicians, 3) at least 4 treatment sessions, in an individual- or group-counseling format, that are greater than 10 minutes in duration, 4) counseling that includes problem-solving, skills training, and social support components, and 5) and the opportunity to use effective medications to aid in tobacco cessation.
  Interventions: Behavioral: Treatment as Usual
- NCI QuitGuide (Active Comparator): Behavioral: The National Cancer Institute's (NCI's) QuitGuide app is a free smartphone app that is available through the Smokefree.gov website. Participants can track cravings, smoking triggers, and motivations for quitting. Participants who are randomly assigned to the QuitGuide app group will receive a smartphone that is preloaded with the QuitGuide app and a quit date scheduled for 1 week after the baseline visit.
  Interventions: Behavioral: QuitGuide
- Smart-T (Experimental): Behavioral: The Smart-Treatment (Smart-T) phone based smoking cessation intervention has multiple components (e.g., an on-demand "Quit Tips" function, an on-demand "Medications" function/button that offers information about nicotine replacement therapy (NRT), button available 24/7 that offers general smoking cessation advice, daily treatment messages, and an algorithm that uses participant's EMA responses to assess risk of lapse and automatically push relevant messages to help them avoid smoking).
  Interventions: Behavioral: Smart-T

INTERVENTIONS:
Behavioral: Treatment as Usual — Tobacco Treatment Research Program (TTRP) or Treatment as Usual (TAU)
  Arms: Treatment as Usual
Behavioral: QuitGuide — NCI QuitGuide Treatment App
  Arms: NCI QuitGuide
Behavioral: Smart-T — Smart-Treatment App
  Arms: Smart-T

SUMMARY:
The primary long-term objective of this research is to reduce smoking relapse through the use of automated mobile smoking cessation interventions that tailor content (e.g., treatment messages/materials) in real-time based upon currently present symptoms. The primary short-term objective of this pilot study is to determine the initial utility of a novel smartphone based smoking cessation intervention compared with standard in-person smoking cessation clinic care and the free National Cancer Institute (NCI) QuitGuide smoking cessation application. The current pilot study is a 3 armed randomized clinical trial that aims to determine the initial utility of a novel smartphone based smoking cessation intervention compared with standard in-person smoking cessation clinic care and the free NCI QuitGuide smoking cessation application.

DETAILED DESCRIPTION:
Description of Study Visits.

Screening and Baseline Assessment (Visit 1). Individuals attending the orientation visit of the Tobacco Treatment Research Clinic (TTRC) will be provided with detailed information about the study and given the opportunity to have their questions answered within a private room to ensure confidentiality. Study staff will review the consent form with interested participants, and they will be screened for eligibility on-site in a private room in the clinic. Participants will be questioned about their 1) age, 2) current level of smoking, 3) willingness to quit smoking, and 4) willingness/ability to attend 4 sessions (including the first visit). Participants will be randomized to treatment as usual (TAU), QuitGuide, or Smart-T groups and advised of their group assignment. Participants will complete the assessment portion of visit 1. Participants will complete self-report questionnaires on a laptop/tablet computer; and weight, and height will be measured in a private room to ensure confidentiality. Participants will be loaned an Android smartphone and instructed regarding the use of the phone as well as the ecological momentary assessment (EMA) procedures.

Quit Day (Visit 2). Participants will complete self-report questionnaires on a laptop/tablet computer; and expired CO and weight will be measured in a private room to ensure confidentiality. Participants will compensated completion of the in-person assessments. All questions about study phones will be appropriately addressed and answered. Participants who do not attend will be contacted by phone to obtain their self-reported smoking status.

4 Weeks Post-Quit (Visit 3). Participants will complete self-report questionnaires on a laptop/tablet computer; and expired CO and weight will be measured in a private room to ensure confidentiality. Participants will be compensated for the completion of the in-person assessments, which will take approximately 45-60 minutes to complete. When participants return the phone they will be compensated according to the compensation schedule described above. Participants who do not attend will be contacted by phone to obtain their self-reported smoking status and to request that the study phone be returned by mail or in-person at the next visit.

12 Weeks Post-Quit (Visit 4; Follow-Up). Participants will complete self-report questionnaires on a laptop/tablet computer; and expired CO and weight will be measured in a private room to ensure confidentiality. Participants will be compensated for the completion of the in-person assessments, which will take approximately 60 minutes to complete. Participants who do not attend will be contacted by phone to obtain their self-reported smoking status.

ELIGIBILITY:
Inclusion Criteria:

1. earn a score ≥ 4 on the Short REALM indicating > 6th grade English literacy level,
2. are willing to quit smoking 7 days from their first visit,
3. are ≥ 18 years of age,
4. have an expired carbon monoxide (CO) level > 7 ppm suggestive of current smoking,
5. are currently smoking ≥ 5 cigarettes per day,
6. are willing and able to attend 4 assessment sessions (i.e., baseline, quit day [1 week after baseline], 4 weeks post-quit, 12 weeks post-quit), and
7. have no contraindications for over the counter NRT (i.e., individuals with uncontrolled blood pressure, history of myocardial infarction within the past two weeks, or current pregnancy, breastfeeding, or plans to become pregnant during the study period will be excluded).

Exclusion Criteria:

1. cannot read, speak, and understand English
2. are < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Biochemically-verified smoking cessation | 12 weeks post-quit
  Biochemically-verified smoking cessation will be verified if the participants have a CO level of < 10 on the quit day and < 6 ppm at all subsequent post-quit visits

CONTACTS AND LOCATIONS:
Overall Officials: Michael Businelle, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center - OTRC, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benson L, Chen M, De La Torre I, Hebert ET, Alexander A, Ra CK, Kendzor DE, Businelle MS. Associations between morning affect and later-day smoking urges and behavior. Psychol Addict Behav. 2024 May;38(3):277-295. doi: 10.1037/adb0000970. Epub 2023 Dec 14. PMID 38095939
- [Derived] Benson L, Ra CK, Hebert ET, Kendzor DE, Oliver JA, Frank-Pearce SG, Neil JM, Businelle MS. Quit Stage and Intervention Type Differences in the Momentary Within-Person Association Between Negative Affect and Smoking Urges. Front Digit Health. 2022 Mar 29;4:864003. doi: 10.3389/fdgth.2022.864003. eCollection 2022. PMID 35425934
- [Derived] Hebert ET, Ra CK, Alexander AC, Helt A, Moisiuc R, Kendzor DE, Vidrine DJ, Funk-Lawler RK, Businelle MS. A Mobile Just-in-Time Adaptive Intervention for Smoking Cessation: Pilot Randomized Controlled Trial. J Med Internet Res. 2020 Mar 9;22(3):e16907. doi: 10.2196/16907. PMID 32149716